CLINICAL TRIAL: NCT07243015
Title: Exosomal microRNA-based Analysis for Early detectIon of Gastric Cancer Hidden-recurrence Traces
Brief Title: Detection of Minimal Residual Disease Using Exosomal miRNA Distant Metastasis Markers
Acronym: ENLIGHT
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/ENLIGHT
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer
Keywords: GC; MRD; Tumor recurrence; Exosomal microRNAs; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Exosomal microRNAs in plasma or serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Discovery Cohort - Distant Metastasis Positive: Patients with postoperative distant metastasis; used for biomarker discovery via small RNA sequencing.
  Interventions: Diagnostic Test: small RNA-seq or array
- Discovery Cohort - Distant Metastasis Negative: Patients without postoperative metastasis; used as reference controls in discovery phase.
  Interventions: Diagnostic Test: small RNA-seq or array
- Training Cohort - MRD Positive (High Risk): Patients exhibiting postoperative recurrence within 12 months.
  Interventions: Diagnostic Test: ENLIGHT Assay
- Training Cohort - MRD Negative (Low Risk): Patients without recurrence ≥12 months postoperatively.
  Interventions: Diagnostic Test: ENLIGHT Assay
- Validation Cohort - MRD Positive: Independent validation cohort with confirmed distant metastasis or MRD positivity.
  Interventions: Diagnostic Test: ENLIGHT Assay
- Validation Cohort - MRD Negative: Independent validation cohort without recurrence/metastasis.
  Interventions: Diagnostic Test: ENLIGHT Assay

INTERVENTIONS:
Diagnostic Test: small RNA-seq or array — small RNA-seq or array
  Groups: Discovery Cohort - Distant Metastasis Negative; Discovery Cohort - Distant Metastasis Positive
Diagnostic Test: ENLIGHT Assay — RT-qPCR-based exo-miRNA quantification
  Groups: Training Cohort - MRD Negative (Low Risk); Training Cohort - MRD Positive (High Risk); Validation Cohort - MRD Negative; Validation Cohort - MRD Positive

SUMMARY:
Gastric cancer (GC) is a leading cause of cancer-related death worldwide. Even in patients undergoing curative surgery for non-metastatic disease, postoperative recurrence frequently occurs due to undetected minimal residual disease (MRD). This study aims to establish a highly sensitive and specific liquid biopsy assay using exosomal microRNAs (exo-miRNAs) to detect MRD and predict distant metastasis before clinical recurrence.

DETAILED DESCRIPTION:
Postoperative recurrence in gastric cancer is largely driven by occult micrometastatic disease that remains undetectable by conventional imaging. While circulating tumor DNA (ctDNA) assays have shown utility in MRD detection, their limited sensitivity and tumor-type variability hinder consistent application in gastric cancer.

Exosomal microRNAs (exo-miRNAs), encapsulated within lipid bilayer vesicles, remain stable in circulation and reflect tumor-derived molecular information. This study seeks to develop and validate an exosomal miRNA-based signature capable of detecting minimal residual disease and predicting future distant metastasis after curative gastrectomy.

Study Phases

1. Discovery Phase - Comprehensive small RNA sequencing to identify miRNAs specific to distant metastasis in gastric cancer.
2. Training Phase - RT-qPCR-based quantification of candidate exo-miRNAs in postoperative plasma samples to develop an MRD signature.
3. Validation Phase - Independent cohort testing to evaluate the diagnostic performance, sensitivity, and specificity of the exosomal MRD panel.

Ultimately, the ENLIGHT assay aims to guide postoperative adjuvant chemotherapy by stratifying patients according to MRD status, enabling precision surveillance and early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma.
* Underwent curative-intent resection (R0).
* Availability of pre- and postoperative plasma samples.
* Documented clinical follow-up data (recurrence/metastasis status).
* Provided written informed consent.

Exclusion Criteria:

* Insufficient plasma volume or RNA quality for exosomal extraction.
* Presence of synchronous or metachronous malignancies.
* Received neoadjuvant chemotherapy without postoperative follow-up.
* Lack of consent or incomplete clinicopathologic data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent curative-intent gastrectomy for gastric adenocarcinoma, with available pre- and postoperative plasma samples.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | up to 5 years
  Time from surgery to recurrence or death.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 5 years
  Time from surgery to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data